CLINICAL TRIAL: NCT01040637
Title: A Phase 1/Phase 2, Randomized, Double-Blind, Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Effect on Opioid Analgesia of TD-1211 Administered Orally to Healthy Volunteers and to Assess the Safety, Pharmacokinetics, and Effect on Bowel Movements in Subjects With Opioid-Induced Constipation
Brief Title: A Multiple Dose Study of TD-1211 in Healthy Volunteers and Patients With Opioid-Induced Constipation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0067
Record Dates: First submitted 2009-12-22; First posted 2009-12-29 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy; Opioid-induced Constipation
Keywords: Healthy subjects
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- TD-1211 dose level 1 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 dose level 2 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 dose level 3 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 dose level 4 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 OIC dose level 1 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 OIC dose level 2 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 OIC dose level 3 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 OIC dose level 4 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- TD-1211 OIC dose level 5 (Experimental): Ascending doses
  Interventions: Drug: TD-1211
- Placebo (Placebo Comparator): Ascending doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-1211 — Dose level 1
  Arms: TD-1211 dose level 1
Drug: TD-1211 — Dose level 2
  Arms: TD-1211 dose level 2
Drug: TD-1211 — Dose level 3
  Arms: TD-1211 dose level 3
Drug: TD-1211 — Dose Level 4
  Arms: TD-1211 dose level 4
Drug: TD-1211 — Ascending doses
  Arms: TD-1211 OIC dose level 1
Drug: TD-1211 — Ascending doses
  Arms: TD-1211 OIC dose level 2
Drug: TD-1211 — Ascending doses
  Arms: TD-1211 OIC dose level 3
Drug: TD-1211 — Ascending doses
  Arms: TD-1211 OIC dose level 4
Drug: TD-1211 — Ascending doses
  Arms: TD-1211 OIC dose level 5
Drug: Placebo — Ascending doses
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of TD-1211 in healthy subjects and activity in subjects with opioid-induced constipation (OIC).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive
* Healthy subjects and subjects with documented OIC on stable opioid regimen
* Willingness to stop all laxatives throughout the OIC screening and treatment period

Exclusion Criteria:

* Any clinically significant finding in healthy subjects
* Have participated in another clinical trial of an investigational drug 30 days prior to screening
* History of chronic constipation prior to opioid therapy in OIC subjects
* Active medical disorders associated with diarrhea or intermittent loose stools in OIC subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in healthy subjects and activity in subjects with opioid-induced constipation | Daily pre and post dose assessments throughout the duration of the study period

SECONDARY OUTCOMES:
Evaluation of the multiple dose pharmacokinetics of TD-1211 following oral administration | Daily pre and post dose assessments throughout the duration of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (3):
- United States (3):
  - Clinical Research Unit, Pasadena, California
  - Clinical Research Unit, San Antonio, Texas
  - Clinical Research Unit, Salt Lake City, Utah